CLINICAL TRIAL: NCT07407322
Title: Effect of Affirmation-Based Information on Stress and Intolerance of Uncertainty in High-Risk Pregnant Women Admitted to the Emergency Department: A Randomized Controlled Trial
Brief Title: Affirmation-Based Information for Stress Reduction in High-Risk Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nilgun Avci (Other)
Responsible Party: Sponsor-Investigator, Nilgun Avci, phD, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Stress Reduction in High-Risk
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: High-risk Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Affirmation-Based Information (Experimental): Pregnant women received routine emergency obstetric care, structured verbal information about the emergency unit and their current condition, followed by affirmation statements delivered verbally in a calm and supportive tone during non-stress test monitoring.
  Interventions: Behavioral: Affirmation + Information Group
- Control group (No Intervention): Pregnant women received routine emergency obstetric care and structured verbal information about the emergency unit and their current condition during non-stress test monitoring.

INTERVENTIONS:
Behavioral: Affirmation + Information Group — Pregnant women received routine emergency obstetric care, structured verbal information about the emergency unit and their current condition, followed by affirmation statements delivered verbally in a calm and supportive tone during non-stress test monitoring.
  Arms: Affirmation-Based Information

SUMMARY:
This study examined whether providing affirmation-based information to high-risk pregnant women admitted to the obstetrics emergency department could reduce stress levels and intolerance of uncertainty. High-risk pregnancy can be emotionally challenging, especially in emergency settings, and supportive communication may help women cope with stress during this period.

In this randomized controlled trial, pregnant women diagnosed with high-risk pregnancy were assigned either to an intervention group that received routine emergency care along with verbal information and positive affirmation statements, or to a control group that received routine emergency care and verbal information only. Stress levels and intolerance of uncertainty were measured before and after the intervention using validated assessment tools.

The findings of this study aim to contribute to evidence-based supportive care practices in obstetric emergency settings and to inform health care professionals about non-pharmacological approaches to improving emotional well-being in high-risk pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Gestational age of 32 weeks or above
* Diagnosed with high-risk pregnancy
* Admitted to the obstetrics emergency department
* Volunteered to participate and provided written informed consent

Exclusion Criteria:

* Inability to communicate in Turkish
* No diagnosis of high-risk pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Level | Baseline and immediately after the intervention during emergency department observation
  Change in perceived stress measured by the Neuman Systems Model-Based Perceived Stress Scale for High-Risk Pregnancy.

SECONDARY OUTCOMES:
Intolerance of Uncertainty | Baseline and immediately after the intervention
  Change in intolerance of uncertainty measured by the Intolerance of Uncertainty Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- State Obstetrics and Gynecology Hospital, Istanbul, Bayrampaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No